CLINICAL TRIAL: NCT06976151
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Dysmenorrhea Among Autoimmune Disease Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lamiaa Mostafa Okeil, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004759
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical treatment group (Active Comparator): The participants will receive non-steroidal anti-inflammatory drugs (NSAID) for 3 consecutive menstrual cycle.
  Interventions: Drug: Non-steroidal anti-inflammatory drugs (NSAID)
- Transcutaneous Electrical Acupoint Stimulation (TEAS) group (Experimental): The participants will receive Transcutaneous Electrical Acupoint Stimulation (TEAS), 3 days per week for 3 consecutive menstrual cycle.
  Interventions: Drug: Non-steroidal anti-inflammatory drugs (NSAID); Other: Transcutaneous Electrical Acupoint Stimulation (TEAS)

INTERVENTIONS:
Drug: Non-steroidal anti-inflammatory drugs (NSAID) — The participants will receive non-steroidal anti- inflammatory drugs (NSAID), Diclofenac 20 mg/ day for 3 consecutive menstrual cycles.
Other: Transcutaneous Electrical Acupoint Stimulation (TEAS) — The participants will receive transcutaneous electrical acupoint Stimulation (TEAS). These acupoints will include large intestine 14 (LI4) , gall bladder 34 (GB34), large intestine 11 (LI11), Gall bladder 39 (GB39) and stomach 36 (ST 36). The session will be applied for 30 minutes / 3 days/ week, in addition to Diclofenac 20 mg/ day for 3 consecutive menstrual cycles.
  .
  Arms: Transcutaneous Electrical Acupoint Stimulation (TEAS) group

SUMMARY:
This study will be conducted to investigate transcutaneous electrical acupoint stimulation effect on pain and disease aggravation during menstruation among autoimmune disease women

DETAILED DESCRIPTION:
The monthly ovarian cycle is characterized by tightly regulated hormones predictably fluctuating throughout the reproductive years. The menstrual cycle plays a role in the exacerbation of rheumatologic conditions, such as rheumatoid arthritis and systemic lupus erythematosus, with flares occurring prior to and during menses, respectively Given these previous observations, sex hormones are hypothesized to influence the biologic properties of the immune system and skin.

Women with rheumatoid arthritis (RA) reported increased pain, fatigue, and disease activity right before their period. Furthermore, those with systemic lupus erythematosus (SLE) experienced similar symptom flares during menses.

The transcutaneous electrical acupoint stimulation (TEAS) is a combination of transcutaneous electrical nerve stimulation (TENS) and traditional Chi- nese acupoints. . Electroacupuncture blocks pain by activating a variety of bioactive chemicals through peripheral, spinal, and supraspinal mechanisms such as the prompt release of β-endorphin and met-enkephalin . Corticotrophin-releasing factor and prostaglandin E2 are also involved in electroacupuncture analgesia.

There are growing literature to support the relationship between the aggravation of autoimmune disease symptoms during menstruation time which maximizes the negative effect on the female's the daily activities at that time. There is lack of researches on the effect of TEAS on this point .TEAS has positive effect on pain during menstrual cycle . The result of this study will help to evaluate the efficacy of TEAS on Pain and disease severity during menstruation in women with autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* All women will be diagnosed with Rheumatoid arthritis(RA) or Systemic lupus erythematosus (SLE).
* All women will suffer from severe pain during menstruation
* Age will range from 25-40 years old.
* Body mass index: 18.5- 30 Kg/m²
* All women participated in the study will have regular menstrual cycle

Exclusion Criteria:

* Secondary dysmenorrhea
* Any other autoimmune diseases not mention in research
* Cardiac or respiratory diseases
* Vaginal infection
* Anemia diseases

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
10 meter walk test | 3 months
  Each woman in both groups will receive the 10 meter walk test to determine functional mobility, gait, and vestibular function.
  Calculating Gait Speed - total distance/time. For example: if you did a 10-meter gait speed test and it took you 7 seconds, the equation would like: 10 meters / 7 seconds = 1.4 meters per second. Normative Values, age 20-29 years : Average Walking Speed(m/s): 1.36-1.34 m/s, age: 30-39 years: Average Walking Speed(m/s):1.43-1.34 m/s.
Assessment of degree of pain | 3 months
  Each woman in both groups will have visual analogue scale (VAS) for conducting of degree of pain in joints just before and during menstruation for 3 consecutive menstruation. It is pointed from 0 to 10 , 0 means no pain and 10 is worst pain
Erythrocyte sedumntation rate (ESR) | 3 months
  It is a type of blood test that measures how quickly erythrocytes (red blood cells) settle at the bottom of a test tube that contains a blood sample. The blood samples will be collected at the beginning and after the end of treatment procedures to detect the level of inflammation for both groups. normal value ranges from 0 to 20 mm/hr.
C-reactive protein (CRP) | 3 months
  It is a substance the liver produces in response to inflammation. The blood samples will be collected at the beginning and after the end of treatment procedures to detect the level of inflammation for both groups. Normal value is less than 0.9 mg/dl.
Pain disability index (PDI) | 3 months
  The Pain Disability Index (PDI) a simple and rapid instrument for measuring the impact that pain has on the ability of a person to participate in essential life activities. I t includes the following items family and home responsibilities, recreation, social activity, occupation, self care, and life-support activity. It is scored from 0 to 10. 0 means no disability and 10 means worst disability.

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Kamel, Professor, Study Director — Cairo University; Amel Youssef, Professor, Study Chair — Cairo University
Locations (1):
- Lamiaa Mostafa Okeil, Al Fayyum, Egypt